CLINICAL TRIAL: NCT01353300
Title: Investigation of DICER1 in Cystic Nephroma and Cystic Partially Differentiated Nephroblastoma
Brief Title: Gene Mutation in Samples From Young Patients With Pleuropulmonary Blastoma Syndrome at Risk for Developing Cancer
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN11B2; COG-AREN11B2 (Other: Children's Oncology Group); NCI-2011-02854 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AREN11B2 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-05-12; First posted 2011-05-13 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Brain and Central Nervous System Tumors; Hereditary Wilms Tumor; Kidney Cancer; Liver Cancer; Neuroblastoma; Pleuropulmonary Blastoma; Sarcoma
Keywords: embryonal childhood rhabdomyosarcoma; cystic nephroma; neuroblastoma; childhood medulloblastoma; childhood hepatoblastoma; stromal predominant Wilms tumor; hereditary Wilms tumor; pleuropulmonary blastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Kidney Neoplasms; Liver Neoplasms; Neuroblastoma; Pleuropulmonary blastoma; Sarcoma; Medulloblastoma; Hepatoblastoma | interventions — Cytogenetic Analysis; Gene Expression Profiling; Gene Rearrangement; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: cytogenetic analysis
Genetic: gene expression analysis
Genetic: gene rearrangement analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: The identification of gene mutations in young patients with pleuropulmonary blastoma syndrome may allow doctors to better understand the genetic processes involved in the development of some types of cancer, and may also help doctors identify patients who are at risk for cancer.

PURPOSE: This research study studies gene mutations in samples from young patients with pleuropulmonary blastoma syndrome at risk for developing cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if DICER1 mutations contribute to tumor pathogenesis in cystic nephromas and cystic partially differentiated nephroblastomas outside of families with pleuropulmonary blastoma (PPB) syndrome.

OUTLINE: Archived DNA samples are analyzed for DICER1 mutation by qPCR and directly sequenced using BigDye Terminator chemistry. Results are then compared against the single nucleotide polymorphism (SNP) database.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of pleuropulmonary blastoma syndrome
* Normal tissue samples, if available
* Parental and sibling DNA samples, if available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of pleuropulmonary blastoma syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2011-05; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Relationship between DICER1 mutations and tumor pathogenesis in cystic nephromas and cystic partially differentiated nephroblastomas outside of families with PPB nephroblastomas

CONTACTS AND LOCATIONS:
Overall Officials: Dana A. Hill, MD, Principal Investigator — Children's National Research Institute